CLINICAL TRIAL: NCT04252924
Title: The Prevalence of Healthy Lifestyle in Students in Europe: the Mediterranean Diet, Orthorexia Nervosa, Appropriate Physical Activity, Stress Perception, and Sleep Habits
Brief Title: Habits, Orthorexia Nervosa and LIfestyle in STudents
Acronym: HOLISTic
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Split, School of Medicine (Other)
Collaborators: University of Pavia (Other); University of Foggia (Other); Beirut Arab University (Other); University of Wroclaw (Unknown); University of Agricultural Sciences and Veterinary Medicine Cluj-Napoca (Unknown); Universidad Pablo de Olavide (Other)
Responsible Party: Principal Investigator, Ivana Kolcic, Associate Professor, University of Split, School of Medicine
Other Study IDs: USplitSM2
Record Dates: First submitted 2020-01-30; First posted 2020-02-05 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: Habits; Health Behavior; Diet Habit; Sleep; Stress; Physical Activity
Keywords: Mediterranean diet; physical activity; sleep; stress; orthorexia nervosa
MeSH Terms: conditions — Habits; Health Behavior; Feeding Behavior; Motor Activity; Orthorexia Nervosa

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- students: medical student, dental medicine student, pharmacy student, nursing student, physiotherapy student, dietetics student, kinesiology student, biomedical laboratory techniques student, biomolecular science student, psychology student, economy student, student of maritime sciences
  Interventions: Other: lifestyle characteristics

INTERVENTIONS:
Other: lifestyle characteristics — Exposures of interest: Mediterranean diet, orthorexia nervosa, smoking, physical activity, sleep duration, stress level

SUMMARY:
Non-communicable diseases (NCDs) compose a substantial proportion of the global burden of diseases, posing a significant challenge in both high-income and low- and middle-income countries. In particular, certain lifestyle-related risk factors, such as unhealthy diet, physical inactivity, smoking, excessive alcohol consumption, and sleep deprivation are the leading risk factors, which place people at an increased risk of developing NCDs. On the other hand, a growing phenomenon of excessive concern about diet and health is emerging, and it is contributing to the development of a novel eating behavior disorder named orthorexia nervosa. According to recent studies, orthorexic behavior is very common among young adults and especially so in health-care professionals.

The main objective of this multi-center study is to explore and compare lifestyle habits among undergraduate medical students and other healthcare-related professions from different countries (Croatia, Lebanon, Italy, Poland, Spain, and Turkey). The goal is to obtain information on the presence of unhealthy habits in order to be able to intervene, offering the information needed for primordial disease prevention in this young and still healthy group of respondents, who are the health educators and role models of the future. The particular importance of this goal is to raise awareness of the problem of the ubiquitously present unhealthy lifestyles. Unfortunately, health-care students are not the exception regarding the prevalence of the unhealthy diet, sedentary behavior, sleep deprivation and high levels of psychological stress. Furthermore, the adoption of unhealthy lifestyle patterns in health-care workers, such as doctors and nurses, will have far-reaching negative consequences, in both their health and their patients' health. The results of this study will be used for identifying the needs and targets for intervention, enabling students to become a pillar of health education for their patients and the population in general.

ELIGIBILITY:
Inclusion Criteria:

1. students enrolled in any of the health-care related studies:

   * medical students
   * dental medicine students
   * pharmacy students
   * nursing students
   * physiotherapy students
   * dietetics/nutrition students
   * biomolecular science students
   * biomedical laboratory techniques students
   * psychology students
2. economy students
3. students of maritime sciences

Exclusion Criteria:

* none

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study population includes the overall student population from the following universities:
  University of Split (Split, Croatia), University of Pavia (Pavia, Italy), University of Foggia (Foggia, Italy), Koc University (Istanbul, Turkey), Beirut Arab University (Beirut, Lebanon), University of Social Sciences and Humanities (Katowice, Poland), University of Agricultural Sciences and Veterinary Medicine Cluj-Napoca (Cluj-Napoca, Romania), Universidad Pablo De Olavide (Sevilla, Spain)
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2018-04-20 (Actual); Primary Completion 2021-04-20 (Estimated); Study Completion 2021-04-20 (Estimated)

PRIMARY OUTCOMES:
the Mediterranean diet adherence | 1 day
  Based on the modern Mediterranean diet pyramid and assessed using the scoring system called Mediterranean Diet Serving Score (MDSS; PubMed ID: 26035442). This score has a minimum value of 0 and a maximum value of 24, where the higher score indicates a better compliance with the Mediterranean diet. Additionally, a cut-off point of 14 and more was proposed to indicate the good adherence to the Mediterranean diet.
moderate to vigorous level of physical activity | 1 day
  Based on self-reported data using a questionnaire called International Physical Activity Questionnaire - Short Form (IPAQ-SF; PubMed ID: 12900694). The MET-min (the metabolic equivalent of task) per week are calculated as: MET level x minutes of activity x events per week. Higher number of MET-min per week denotes higher level of physical activity (a better outcome). Details on the scoring protocol can be found at: https://sites.google.com/site/theipaq/scoring-protocol
sleep duration | 1 day
  Based on self-reported data using a questionnaire (time of going to sleep and waking up)
stress level | 1 day
  Based on self-reported data using a questionnaire called Perceived Stress Scale (PSS; PubMed ID: 6668417). The scale has a minimum score of 0 and a maximum of 40, where higher score indicates higher perceived stress during last month.

SECONDARY OUTCOMES:
Orthorexia nervosa | 1 day
  Based on self-reported data using the questionnaire the Eating Habits Questionnaire (EHQ). The scale has a minimum score of 21, and a maximum score of 84, where higher score indicates higher orthorexic symptoms. Additionally, the scale has three sub scales: knowledge of healthy eating, problems associated with healthy eating, and feeling positively about healthy eating.
Orthorexia nervosa | 1 day
  Based on self-reported data using the Orthorexia nervosa questionnaire (ORTO-15; PubMed ID: 16682853). ORTO-15 has a minimum score of 15 and a maximum of 60, where lower score denotes higher orthorexic symptoms, and the cut-off value of <40 has been proposed to indicate higher probability for the presence of orthorexia.

CONTACTS AND LOCATIONS:
Overall Officials: Ivana Kolcic, Assoc. Prof., Principal Investigator — University of Split, School of Medicine
Locations (8):
- Ivana Kolcic, Split, Croatia
- Italy (2):
  - Department of Economics, University of Foggia, Foggia
  - University of Pavia, Pavia
- Beirut Arab University, Beirut, Lebanon
- Institute of Psychology, University of Wroclaw; University of Social Sciences and Humanities (Katowice), Wroclaw, Poland
- Faculty of Veterinary Medicine, University of Agricultural Sciences and Veterinary Medicine, Cluj-Napoca, Romania
- Universidad Pablo De Olavide, Seville, Spain
- Koc University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
Depends upon the agreement of all study sites investigators

REFERENCES:
- [Background] Monteagudo C, Mariscal-Arcas M, Rivas A, Lorenzo-Tovar ML, Tur JA, Olea-Serrano F. Proposal of a Mediterranean Diet Serving Score. PLoS One. 2015 Jun 2;10(6):e0128594. doi: 10.1371/journal.pone.0128594. eCollection 2015. PMID 26035442
- [Background] Craig CL, Marshall AL, Sjostrom M, Bauman AE, Booth ML, Ainsworth BE, Pratt M, Ekelund U, Yngve A, Sallis JF, Oja P. International physical activity questionnaire: 12-country reliability and validity. Med Sci Sports Exerc. 2003 Aug;35(8):1381-95. doi: 10.1249/01.MSS.0000078924.61453.FB. PMID 12900694
- [Background] Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983 Dec;24(4):385-96. No abstract available. PMID 6668417
- [Background] Gleaves DH, Graham EC, Ambwani S. Measuring 'Orthorexia': Development of the Eating Habits Questionnaire. International Journal of Educational and Psychological Assessment. 12(2):1-18, 2013.
- [Background] Donini LM, Marsili D, Graziani MP, Imbriale M, Cannella C. Orthorexia nervosa: validation of a diagnosis questionnaire. Eat Weight Disord. 2005 Jun;10(2):e28-32. doi: 10.1007/BF03327537. PMID 16682853